CLINICAL TRIAL: NCT00369759
Title: An Epidemiological Study to Evaluate the Seasonality of Respiratory Syncytial Virus-Associated-Lower Respiratory Tract Infections (LRI) or Apnea in Infants in the Emergency Department
Brief Title: An Epidemiological Study to Evaluate the RSV-Associated Lower Respiratory Track in Infections in Infants
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Responsible Party: Jessie Groothuis, MD, MedImmune Inc.
Other Study IDs: MI-MA133
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Respiratory Infections; Bronchiolitis; Pneumonia; Apnea
Keywords: Acute Lower Respiratory Infection; Retractions; Bronchiolitis or pneumonia; Wheezing; Rales; Crackles
MeSH Terms: conditions — Respiratory Tract Infections; Bronchiolitis; Pneumonia; Apnea; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal wash specimen (RSV)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Bronchiolitis, pneumonia or Lower Respiratory Infection or LRI (Season 1: 2006-'07 and same for Season 2: 2007 - '08)
  Interventions: Other: Emergency Dept. Subjects with LRI or Apnea
- 2: Bronchiolitis, pneumonia or Lower Respiratory Infection or LRI (Season 1: 2006-'07 and same for Season 2: 2007 - '08)
  Interventions: Other: Emergency Dept. Subjects with LRI or Apnea
- 3: Bronchiolitis, pneumonia or Lower Respiratory Infection or LRI (Season 1: 2006-'07 and same for Season 2: 2007 - '08)
  Interventions: Other: Emergency Dept. Subjects with LRI or Apnea

INTERVENTIONS:
Other: Emergency Dept. Subjects with LRI or Apnea — No intervention; Epidemiological Study

SUMMARY:
The primary objective of this study is to describe the incidence of RSV-associated LRI among infants <1 year of age presenting to the ED during selected shoulder months.

DETAILED DESCRIPTION:
* The primary objective of this study is to describe the incidence of RSV-associated LRI or apnea (% RSV positive) among infants <1 year of age presenting to the ED during selected shoulder months. The total number of events will also be described.
* To characterize the clinical outcomes and demographic data of infants presenting to the ED with RSV-associated LRI or apnea
* To characterize the social burden (in the form of number of days lost from work by parent/ guardian) for these infants through 14 days after the index ED visit and through hospital discharge will also be described.
* Based on a sample of cases collected in a cohort of patients enrolled at or near the peak of RSV disease during the traditional season, a comparison of the rate of RSV between shoulder and peak periods will be described.
* To describe the overall rates of RSV-associated LRI or apnea based on the general ED statistics collected during the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from parent/guardian to participate in this study
* Male and female infants <1 year of age (child must be entered before his/her 1st birthday)
* Physician diagnosis of either a) acute LRI or b) apnea below:

A) Acute LRI, defined as:

1. Medical diagnosis of bronchiolitis or pneumonia, or
2. In the absence of either of these diagnoses, LRI will be determined by the investigator after review of the medical record and must include at least one of the following:

   * Retractions
   * Wheezing
   * Rales or crackles
   * The presence of a new infiltrate, if a chest X-ray is available, which must be diagnosed by the ED physician or radiologist

B) Apnea, defined as either:

1. Cessation of breathing for >20 seconds by history or observation, or
2. Cessation of breathing for any length of time if accompanied by cyanosis or pallor, bradycardia as detected by a monitor, or
3. ED primary diagnosis of apnea

   * Parent/guardian has the ability and willingness to be available for a follow-up interview by telephone

Exclusion Criteria:

* Use of palivizumab or RSV-IGIV at any time prior to enrollment
* Participation in trials of investigational RSV prophylaxis or therapeutic agents

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible subjects with RSV results.
Sampling Method: Non-Probability Sample
Enrollment: 2048 (Actual)
Dates: Start 2006-09; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Measuring the incidence of RSV-associated, LRI or apnea among infants <1 yr. old presenting the Emergency Dept. during shoulder months. | July 2008

SECONDARY OUTCOMES:
Clinical outcome of infants at Emergency Dept. with RSV-associated LRI or apnea.(hospital admission, 23 hr.-observations,no. of outpatient and/or urgent care visits,ICU,mechanical ventilation,supplemental oxygen use, meds,admission rate) | July 2008
Societal burden(no. of days lost from work by parent/guardian) for infants through 14 days after index ED visit and through hospital discharge. | July 2008
Comparison of rates of RSV-associated LRI or apnea during the peak periods and between shoulder and peak periods. | July 2008
Overall rates of RSV-associated LRI or apnea based on general ED statistics collected during the entire study period, including outside recruitment periods. | July 2008

CONTACTS AND LOCATIONS:
Overall Officials: Jessie R. Groothuis, M.D., Study Director — MedImmune LLC
Locations (37):
- United States (37):
  - Maricopa Medical Center, Phoenix, Arizona
  - Olive View- UCLA Medical Center, Sylmar, California
  - The Children's Hospital, Denver, Colorado
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Alfred J. Dupont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Batchelor Children's Institute, Miami, Florida
  - Miami Children's Hospital Research Institute, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Kentucky Chandler Medical Center/University of Kentucky Clinical Research, Lexington, Kentucky
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Children's National Medical Center, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi, Jackson, Mississippi
  - St. Louis Children's Hospital (Washington University), St Louis, Missouri
  - University of Nebraska Medical Center combined Divistion of Pediatric Infectious Disease, Omaha, Nebraska
  - Children's Hospital of Buffalo, Buffalo, New York
  - Upstate Medical University, Syracuse, New York
  - Wake Forest University Medical Center, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Columbus Children's Hospital - Nationwide Children's of Colombus, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - Doernbecher Children's Hospital Oregon Health Sciences University Hospital, Portland, Oregon
  - Temple University Children's Medical Center, Philadelphia, Pennsylvania
  - Medical University of SC, Charleston, South Carolina
  - University of Tennesee, LeBonheur Children's Med. Center, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas, Southwestern Medical Center, Dallas, Texas
  - Austin Children's Hospital, Temple, Texas
  - Seattle Children's Hospital and Regional Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin